CLINICAL TRIAL: NCT06373406
Title: A Phase I/II, Dose Escalation and Dose Expansion Study of MHB036C for Advanced Solid Tumor to Evaluate the Tolerability/Safety, Pharmacokinetics and Efficacy
Brief Title: A Study of MHB036C for Advanced Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB036C-CP001CN
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB036C (Experimental): MHB036C IV every 3 weeks
  Interventions: Drug: MHB036C

INTERVENTIONS:
Drug: MHB036C — An antibody-drug conjugate therapy

SUMMARY:
Phase I/II, dose escalation and dose expansion study to evaluate the efficacy and safety of MHB036C in advanced malignant tumors.

DETAILED DESCRIPTION:
This first-in-human, dose escalation and dose expansion study is to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of MHB036C in patients with advanced solid tumor. The Phase I stage is to determine the maximum tolerated dose (MTD). The phase II stage is to determine the recommended Phase 2 dose (RP2D) according to safety and efficacy in specific tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily agree to participate in the study and sign the Informed Consent Form (ICF).
* Participants aged 18 years or older (inclusive), without gender limitation.
* Participants with Eastern Cooperative Oncology Group performance score of 0-1.
* Participants with expected survival time of more than 3 months.
* Eligible participants of childbearing potential (males and females) must agree to take reliable contraceptive measures (hormone or barrier method, or absolute abstinence, etc.) with their partners during the study and within at least 90 days after the last dose; female participants of childbearing potential must have a negative results of blood pregnancy test within 7 days before the first dose of the investigational product, and must be non-lactating.
* Participants who are able to understand study requirements, and willing and able to comply with arrangements of study and follow-up procedures.
* Participants to be enrolled in part one must have histologically or cytologically confirmed advanced or metastatic solid tumors, which have failed or are intolerant to standard of care (SOC), or for which no SOC is available;

Exclusion Criteria:

* Participants with 2 or more malignancies (except effectively treated non-melanoma skin cancer, cervical carcinoma in situ or other tumors, or malignancies considered cured) within 5 years prior to sign the Informed Consent Form.
* Participants who have received chemotherapy within 3 weeks prior to the first dose of investigational product, or have received anti-tumor therapy including radiation therapy, biologic therapy, endocrine therapy, immunotherapy, etc. within 4 weeks prior to the first dose; or participants with the following conditions:

  * Medication of nitrosourea or mitomycin C within 6 weeks prior to the first dose of MHB036C;
  * Medication of oral fluoropyrimidines or small molecule targeted agents within 5 half-lives of such drug before first dose of investigational product.
  * Medication of traditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first dose of investigational product.
* Medication of other disapproved investigational products or therapies within 4 weeks prior to the first dose of investigational product.
* Presence of brain metastases and/or carcinomatous meningitis. Participants previously treated for brain metastases may be considered to be enrolled in this study, provided they have been in stable condition for at least 4 weeks, no evidence of new or enlarging brain metastases, or without steroid therapy within 14 days prior to the first dose of investigational product. This exception does not include carcinomatous meningitis, which should be excluded regardless of clinical stability.
* Participants previously received same targeted therapy will be excluded.
* Participants with adverse reactions from previous anti-tumor therapy that have not recovered to ≤Grade 1 as per CTCAE 5.0 (except for toxicities without safety risks as determined by the investigator, such as alopecia, hypothyroidism stably managed by hormone replacement therapy, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with adverse events (AE) | Until 30 days after last dose of MHB036C
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities related to MHB036C which meet pre-defined severity criteria and occurs within the first cycle of treatment

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Until 30 days after last dose of MHB036C
  To analysis the serum concentrations at different timepoints to determine the Cmax
The area under the plasma concentration-time curve (AUC) | Until 30 days after last dose of MHB036C
  To analysis the serum concentrations at different timepoints to determine the AUC
To detectable anti-drug antibodies with treated subjects | Until 30 days after last dose of MHB036C
  The immunogenicity of MHB036C will be assessed by the number of subjects who produce anti-drug antibodies (ADAs)
Objective response rate (ORR) | Until 30 days after last dose of MHB036C
  The ORR is defined as the proportion of subjects with confirmed complete remission (CR) or confirmed partial response (PR), based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China